CLINICAL TRIAL: NCT00219037
Title: A 12 Month, Randomized, Open-label, Multicenter, Study to Assess the Long Term Safety of Aliskiren 150 mg Alone and 300 mg Alone or With the Optional Addition of Hydrochlorothiazide (12.5 mg or 25 mg) in Patients With Essential Hypertension.
Brief Title: Long Term Safety of Aliskiren Alone or With the Optional Addition of Hydrochlorothiazide in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSPP100A2302
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: Hypertension, blood pressure, aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
Assess the long-term safety and tolerability of aliskiren, with the optional addition of HCTZ, in patients with essential hypertension, to ensure long term blood pressure control and protect against end organ damage.

ELIGIBILITY:
Inclusion Criteria

1. Patients with essential hypertension.
2. Patients who are eligible and able to participate in the study.

Exclusion Criteria

1. Severe hypertension.
2. History or evidence of a secondary form of hypertension.
3. History of hypertensive encephalopathy or cerebrovascular accident. Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1955 (Actual)
Dates: Start 2004-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory abnormalities, serious adverse events

SECONDARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 12 months
Change from baseline in mean sitting systolic blood pressure after 12 months
Change from baseline in standing systolic blood and diastolic pressure after 12 months
Diastolic blood pressure less than 90 mmHg or reduction of 10 mmHg or greater from baseline
Blood pressure less than 140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Sites, Germany

REFERENCES:
- [Derived] Sica D, Gradman AH, Lederballe O, Kolloch RE, Zhang J, Keefe DL. Long-term safety and tolerability of the oral direct renin inhibitor aliskiren with optional add-on hydrochlorothiazide in patients with hypertension: a randomized, open-label, parallel-group, multicentre, dose-escalation study with an extension phase. Clin Drug Investig. 2011 Dec 1;31(12):825-37. doi: 10.1007/BF03256921. PMID 22035463